CLINICAL TRIAL: NCT07113171
Title: Comparison of Video Laryngoscopy Versus Conventional Laryngoscopy in Anticipated Difficult Intubation in Patients Undergoing Thyroid Surgery
Brief Title: Comparison of Video Laryngoscopy and Conventional Laryngoscopy for Safe Intubation in Adult Thyroid Surgery Patients With Anticipated Difficult Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Kainat usman, Principal Investigator, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sheikh ZMC/H2
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Difficult Airway Intubation; Airway Management During Operative Procedure
Keywords: Airway Management in Thyroid Surgery; Endotracheal Intubation Techniques; Video Laryngoscopy; Direct Laryngoscopy; Anesthesia in Thyroid Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Conventional Laryngoscopy (Active Comparator): Received endotracheal intubation using conventional direct laryngoscope with a Macintosh blade, performed under general anesthesia in patients undergoing thyroid surgery.
  Interventions: Device: Conventional Direct Laryngoscope
- Group B - Video Laryngoscopy (Experimental): Received endotracheal intubation using video laryngoscope under general anesthesia in patients undergoing thyroid surgery.
  Interventions: Device: Video Laryngoscope

INTERVENTIONS:
Device: Conventional Direct Laryngoscope — The Macintosh laryngoscope blade was used for intubation. The technique involved neck extension to create a direct line of sight to the vocal cords for successful tracheal tube placement.
  Other Names: Direct Laryngoscope
  Arms: Group A - Conventional Laryngoscopy
Device: Video Laryngoscope — The video laryngoscope allowed visualization of the glottis on a monitor without the need for cervical extension, facilitating intubation in anticipated difficult airway cases.
  Other Names: Indirect Laryngoscope
  Arms: Group B - Video Laryngoscopy

SUMMARY:
This clinical study is designed to compare two different techniques used for inserting a breathing tube (a process known as intubation) in adult patients undergoing thyroid surgery who are predicted to have a difficult airway. A difficult airway refers to a situation where it may be challenging to place the breathing tube due to specific anatomical or physical factors such as restricted neck movement, enlarged thyroid gland (goiter), reduced mouth opening, short neck, or increased soft tissue around the neck. The two techniques being assessed are conventional direct laryngoscopy, which is the traditional method requiring neck extension for a direct view of the windpipe, and video laryngoscopy, a modern approach that uses a camera to visualize the vocal cords on a screen with less need for neck manipulation.

In this randomized controlled trial, a total of 60 patients meeting the eligibility criteria will be included and randomly assigned into two equal groups. One group will undergo intubation using the conventional laryngoscope, while the other group will be intubated using the video laryngoscope. The primary aim of this research is to evaluate which method provides a higher success rate of placing the endotracheal tube correctly on the first attempt. Additional outcomes that will be assessed include the total time taken for intubation, whether the intubation was ultimately successful regardless of the number of attempts, and the occurrence of any immediate injuries within the mouth or throat area during or after the procedure.

The underlying hypothesis of the study is that video laryngoscopy will result in a significantly higher first-attempt intubation success rate as compared to conventional laryngoscopy in patients with predicted difficult airways. This study intends to provide clinically useful evidence to guide anesthesiologists in selecting the most effective and safe intubation technique for patients undergoing thyroid surgery, with the goal of minimizing complications and improving procedural outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 60 years
* Both genders will be included
* Patients requiring endotracheal intubation under general anaesthesia for thyroid surgery.
* Patients with anticipated difficult intubation based on the preoperative airway assessment.
* Patients having ASA (American College of Anaesthesiologists) class 1 to 2.

Exclusion Criteria:

* Patients having neck injury
* Patients having cervical spondylopathy
* Patients requiring urgent/ emergency thyroid surgery
* Patients with existing oropharyngeal or laryngeal abnormalities.
* Patients with a history of severe cardiovascular or respiratory diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-18 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-05-18 (Actual)

PRIMARY OUTCOMES:
First-Attempt Intubation Success Rate | During intubation at the time of induction of anesthesia (Day 0, intraoperative)
  Successful placement of the endotracheal tube through the vocal cords into the trachea on the first attempt, confirmed by bilateral chest auscultation and capnography.

SECONDARY OUTCOMES:
Overall Intubation Success Rate | During intubation at the time of induction of anesthesia (Day 0, intraoperative)
  Successful tracheal intubation irrespective of the number of attempts required, verified by standard clinical confirmation methods (auscultation and capnography).
Intubation Time | During intubation at the time of induction of anesthesia (Day 0, intraoperative)
  The time taken from the insertion of the laryngoscope blade between the teeth to confirmation of successful tracheal tube placement. Measured in seconds using a stopwatch. This outcome reflects procedural efficiency between the two techniques.
Incidence of Immediate Oropharyngeal Injuries | Immediately post-intubation (within 5 minutes of tube placement, intraoperative)
  Presence or absence of visible soft tissue trauma, bleeding, or other oropharyngeal injuries observed immediately after intubation through visual inspection by the anesthesiologist.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Irfan Jamil, Principal Investigator — Sheikh Zayed Medical college/Hospital, Rahimyar Khan
Locations (1):
- Sheikh Zayed Medical college/hospital, Rahim Yar Khan, Punjab Province, Pakistan